CLINICAL TRIAL: NCT03969823
Title: Whole Genomic Landscape of EGFR Mutation-Positive Advanced Non-Small Cell Lung Cancer Treated With First-Line Osimertinib (WARRIOR)
Brief Title: Whole Genomic Landscape of Advanced EGFR-mutant NSCLC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ESR-18-14174
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: NSCLC; Osimertinib; EGFR exon 19 deletion or L858R mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib (Experimental): Osimertinib at 80mg dose will be administered orally once daily.
  Interventions: Drug: Tagrisso

INTERVENTIONS:
Drug: Tagrisso — Osimertinib 80mg once daily until disease progression
  Other Names: Osimertinib

SUMMARY:
This is a phase 2 single-arm, non-randomized multicentre and tissue acquisition study to evaluate acquired resistance mechanisms, efficacy, and safety in advanced, EGFR tyrosine kinase inhibitor-naïve NSCLC patients with EGFR-activating mutations who receive a first-line osimertinib orally at a dose of 80mg once daily.

DETAILED DESCRIPTION:
This open-label, single-arm, non-randomized phase 2 exploratory study has been designed to evaluate the mechanisms of resistance to first-line osimertinib 80mg once daily in NSCLC patients with EGFR-activating mutation who were naïve to chemotherapy as well as EGFR TKIs. Acquired resistance to first-line osimertinib is mediated by heterogeneous mechanisms including MET amplification (15%), secondary EGFR mutation including C797S or S768I (7%), PIK3CA mutation (7%), CDK4/6 amplification (5%), KRAS mutation (3%), BRAF mutation (3%), CCND1-3 amplification (3%), CCNE1 amplification (2%), HER2 amplification (2%), and SPTBN1-ALK fusion (1%) using plasma genotyping of FLAURA study (N=91). Therefore, this study is necessary to evaluate resistance mechanisms of ≥1% to first-line osimertinib in NSCLC patients with EGFR-activating mutations using whole-genomic profiling of tumours at pre-treatment and progression which acquisitions are mandatory.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female must be > 19 years of age
3. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
4. Male subjects should be willing to use barrier contraception (see Restrictions, Section 3.8)
5. Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy with local confirmation of the presence of EGFR TKI-sensitizing mutation (EGFR exon 19 deletion or L858R mutation), either alone or in combination with other EGFR mutations excluding EGFR exon 20 insertion mutation
6. Mandatory provision of fresh tumor sample before osimertinib via a biopsy or surgical resection
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Patients must have a life expectancy ≥ 12 weeks.
9. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements
10. Provision of informed consent for whole-genome and whole-exome sequencings

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study
2. Previous treatment with an EGFR TKI
3. Patients with different kinds of cancers within 5 years or with malignants simultaneously (except completely cured skin basal cell carcinoma or uterine cervical cancer)
4. Treatment with an investigational drug within five half-lives or 3 months. Patients receiving an radiotherapy targeting brain metastasis or spinal cord compression within 2 weeks before the beginning of study treatment, receiving an wide field radiotherapy over 30% of spinal cord reactivity or who are unrecovered from radiotherapy toxicity
5. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 weeks prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4
6. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2, prior platinum-therapy-related neuropathy
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required
8. Patients with spinal cord compression, symptomatic or unstable brain metastases except for those patients who have completed definitive therapy and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients who may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic are eligible
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib
10. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
11. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
12. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values: absolute neutrophil count <1.5 x 109/L; platelet count <100 x 109/L; haemoglobin <90 g/L; alanine aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases; serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
13. History of hypersensitivity to any of the active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
14. Patients who are pregnant or breast-feeding
15. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
16. Previous allogeneic bone marrow transplant
17. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of acquired resistance mechanisms to osimertinib at disease progression | Through study completion, an average of 2 years
  Disease progression as defined by investigator assessments according to RECIST1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 2 years
  AEs/SAEs as defined by NCI CTCAE version 5.0
Progression-Free Survival (PFS) | Through study completion, an average of 2 years
  PFS as defined as the time from the date of initiation until the date of first documented progression
Overall Survival (OS) | Through study completion, an average of 2 years
  OS as defined as the time from the date of first dose until death due to any cause
Objective Response Rate (ORR) | Through study completion, an average of 2 years
  ORR using investigator assessments according RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Borame Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No